CLINICAL TRIAL: NCT00545948
Title: Phase II Prospective Study Evaluating the Role of Directed Cisplatin Based Chemo With Either Vinorelbine or Pemetrexed for the Adj Tx of Early Stage NSCLC in Patients Using Genomic Expression Profiles of Chemo Sensitivity to Guide Therapy
Brief Title: Adjuvant Cisplatin With Either Genomic-Guided Vinorelbine or Pemetrexed for Early Stage Non-Small-Cell Lung Cancer
Acronym: TOP0703
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to reproducibility issues with genomics prediction model.
Sponsor: Duke University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000657
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung Cancer; NSCLC; Non-Squamous; Genomics; Guided Therapy; Directed Therapy; Genomic Expression Profiles; Chemotherapy Sensitivity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A-Vinorelbine (Other): Resected tumor was used for genomic expression profiling. Patients with a genomic expression pattern suggestive of vinorelbine sensitivity were given cisplatin + vinorelbine.
  Interventions: Drug: Vinorelbine followed by Cisplatin
- Arm B-Pemetrexed (Other): Resected tumor was used for genomic expression profiling. Patients with a genomic expression pattern suggestive of pemetrexed sensitivity were given cisplatin + pemetrexed.
  Interventions: Drug: Pemetrexed followed by Cisplatin

INTERVENTIONS:
Drug: Vinorelbine followed by Cisplatin — Vinorelbine 25 mg/m2 IV over 6-10 minutes on days 1 and 8, followed by Cisplatin 75 mg/m2 IV over 60 minutes on day 1 (every 21 days x 4 cycles).
  Other Names: Navelbine; Platinol
  Arms: Arm A-Vinorelbine
Drug: Pemetrexed followed by Cisplatin — Pemetrexed 500 mg/m2 IV infusion over approximately 10 minutes on day 1, followed by Cisplatin 75 mg/m2 IV over 60 min on day 1 (every 21 days x 4 cycles)
  Other Names: Alimta; Platinol
  Arms: Arm B-Pemetrexed

SUMMARY:
This study assigned subjects to either cisplatin/vinorelbine or cisplatin/pemetrexed chemotherapy using a genomic based expression profile to determine chemotherapy sensitivity in completely resected early stage non-squamous non-small-cell lung cancer (NSCLC). The vinorelbine-sensitive tumors group received Vinorelbine followed by cisplatin, while the pemetrexed-sensitive tumors group received pemetrexed followed by cisplatin. The primary objective of this trial was to determine whether genomic-based adjuvant chemotherapy treatment increased the 2-year progression-free survival rate in completely resected patients with NSCLC compared to historic controls. Secondary objectives included: 1) estimation of the percentage of completely resected NSCLC tumors that can be adequately analyzed and used to direct specific adjuvant chemotherapy; 2) estimation of the proportion of patients who are assigned to treatment with vinorelbine and pemetrexed; 3) evaluation of drug sensitivity patterns of cisplatin and pemetrexed in both treatment arms; 4) description of the overall median survival experience of treated patients; and 5) assessment of patient understanding and perceptions of participating in a clinical trial evaluating cancer genomics for adjuvant treatment of early stage lung cancer.

DETAILED DESCRIPTION:
The proposed study is a multi-center open label phase II study of the chemotherapy doublets cisplatin/vinorelbine and cisplatin/pemetrexed as adjuvant therapy in early stage non-squamous NSCLC.

Eligible patients had no previous treatment for the current diagnosis of NSCLC. The two treatment groups of patients will be determined by gene expression profile analysis of each patient's tumor: one group of vinorelbine-sensitive patients and one group of pemetrexed-sensitive patients. The genomic expression profiling that was utilized generated a percentage for likelihood of chemotherapy sensitivity. Patients were directed to receive the chemotherapy regimen for which the percentage of predicted sensitivity is highest. For instance, if the model predicted the likelihood of tumor sensitivity was 46% to vinorelbine and 48% to pemetrexed, then the adjuvant chemotherapy would be directed to cisplatin/pemetrexed. Patients whose tumors could not be adequately analyzed for gene expression were offered adjuvant therapy off protocol as deemed appropriate by their primary oncologist. Patients with either squamous or non-squamous cell histology were eligible to participate in this study as indicated in study protocols dated prior to January 25, 2010. An amendment to the protocol on January 25, 2010 indicated inclusion of only non-squamous histology. However, because of low accrual after January 25, 2010 (5 patients, including 2 screen failures), this report reflects the original study outcomes that includes both squamous and non-squamous histologies.

Thirty-one patients with stage IB (> 4 cm), II or IIIA non-squamous NSCLC were enrolled, from which 24 were assigned treatment. The vinorelbine-sensitive tumors group received Vinorelbine 25 mg/m2 days 1 and 8, followed by cisplatin 75 mg/m2 day 1, every 21 days for 4 cycles. The pemetrexed-sensitive tumors group received pemetrexed 500 mg/m2 day 1 followed by cisplatin 75 mg/m2 day 1, every 21 days for 4 cycles. Standard pre-medication regimens included dexamethasone, vitamin B12 and folate supplementation in the pemetrexed group. Patients in both groups will receive up to a maximum of 4 cycles of therapy.

Subsequent reevaluation of the genomic signatures of chemotherapy sensitivity have shown that they were irreproducible, suggesting inaccurate patient assignments into the two treatment arms. As a result, it would be inappropriate to separately analyze outcomes for the different treatment groups. Instead, information from both arms will be combined to reflect the overall measure of two-year progression-free survival in this study. Similarly for secondary objectives, both arms will be combined to address endpoints.

To assess patient understanding and perceptions of participating in a clinical trial evaluating cancer genomics for adjuvant treatment of early stage lung cancer, patients provided responses for the following questions at baseline:

1. Did your doctor talk to you today about choosing chemotherapy treatment for lung cancer based on the genomics of your tumor?
2. How well did you understand what you doctor told you about choosing chemotherapy based on the genomics of your tumor? (circle a number between 1 and 7, where 1 = very poorly and 7 = very well)
3. Do you think the type of chemotherapy that you will get is based on the genomics of your tumor?
4. Do you think you will get better medical care for the treatment of your lung cancer if it is based on the genomics of your tumor?
5. To what extent do you think treating lung cancer based on the genomics of the tumor will lead to more successful treatment strategies? (circle a number between 1 and 7, where 1 = definitely will not lead to a more successful treatment and 7 = definitely will lead to a more successful treatment)
6. How effective do you think chemotherapy will be at stopping your cancer from coming back? (circle a number between 1 and 7, where 1 = not at all effective and 7 = completely effective)
7. To what extent is YOUR lung cancer primarily caused by genetics? (circle a number between 1 and 7, where 1 = not at all caused by genetics and 7 = completely caused by genetics)
8. To what extent to do you think your lung cancer is treatable? (circle a number between 1 and 7, where 1 = definitely not treatable and 7 = definitely treatable)
9. Did your doctor talk to you about your chance of your lung cancer coming back? (Yes - go to question 10, No - go to question 11, Do not know - go to question 11)
10. What did your doctor say was your chance of your cancer coming back? (Low Risk, Moderate or intermediate risk, High risk, Do not know)
11. What do you think is your chance of your lung cancer coming back in the next year on a scale from 1 to 7 where 1=definitely will not come back and 7=definitely will come back?
12. How worried are you that your lung cancer will come back in the next year? (circle a number between 1 and 7, where 1=not at all worried and 7=extremely worried)

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they meet all of the following criteria:

1. Patients with completely resected stage IB (> 4 cm), II, or IIIA Non-Squamous NSCLC. Patient must be enrolled and begin therapy within 4 to 12 weeks from the date of complete surgical resection.
2. Fresh tissue must be available for genomics expression profiling.
3. ECOG performance status of 0 or 1.
4. NO prior chemotherapy, radiation therapy, or biologic/targeted therapy within the last 5 years. Prior therapy with low dose methotrexate or similar medications is allowed if therapy used to treat non-malignant conditions.
5. Age ≥ 18 years.
6. No previous or concomitant malignancy in the past 5 years other than curatively-treated carcinoma in situ of the cervix, or basal cell or squamous cell carcinoma of the skin.
7. No other serious medical or psychiatric illness.
8. Signed informed consent.
9. Required laboratory data within one week of enrollment:

   * ANC or AGC ≥ 1500 per uL;
   * Platelets ≥ 100,000 per uL;
   * Total bilirubin ≤ 1.5 mg/dL;
   * Creatinine ≤ 2 mg/dL; creatinine clearance ≥ 45 mL/min;
   * SGOT/SGPT ≤ 1.5x ULN.
10. Females of child-bearing potential (not surgically sterilized and between menarche and 1 year post menopause) must test negative for pregnancy within 7 days prior to or at the time of enrollment based on a serum pregnancy test. Both sexually active males and females of reproductive potential must agree to use a reliable method of birth control, as determined by the patient and their health care team, during the study and for 3 months following the last dose of study drug.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
2. Concurrent administration of any other anti-tumor therapy (see #4 inclusion for exceptions).
3. Inability to comply with protocol or study procedures.
4. Active infection requiring IV antibiotics, antifungal or antiviral agents, that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
5. Major surgery (other than definitive lung cancer surgery) within two weeks of study or other serious concomitant systemic disorders that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
6. Myocardial infarction having occurred less than 6 months before inclusion, any known uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia, or cardiac failure not controlled by medications.
7. Contraindication to corticosteroids.
8. Inability or unwillingness to take folic acid or vitamin B12 supplementation.
9. Unwillingness to stop taking herbal supplements while on study.
10. Presence of clinically significant third-space fluid collections (for example, ascites or pleural effusions) that cannot be controlled by drainage or other procedures prior to study entry and throughout study enrollment as the distribution of pemetrexed in this fluid space is not fully understood.
11. Inability to discontinue administration of aspirin at a dose > 1300 mg/day or other long acting, non-steroidal anti-inflammatory agents for 2 days before, the day of, and 2 days after the dose of pemetrexed (5 days prior for long-acting agents such as piroxicam). Moderate dose ibuprofen may be continued.
12. Female patients that are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, Ph.D., M.D., Principal Investigator — Duke University Medical Center, Hematology/Oncology, Duke Cancer Institute
Locations (13):
- United States (13):
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Presbyterian HealthCare, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Scotland HealthCare System (Scotland Memorial Hospital), Laurinburg, North Carolina
  - Southeastern Regional Medical Center, Gibson Cancer Center, Lumberton, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Johnston Memorial Hospital Authority, Smithfield, North Carolina
  - Columbus County Hospital, Whiteville, North Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Coastal Cancer Center, Myrtle Beach, South Carolina
  - Community Memorial Health Center, South Hill, Virginia

REFERENCES:
- [Background] Potti A, Mukherjee S, Petersen R, Dressman HK, Bild A, Koontz J, Kratzke R, Watson MA, Kelley M, Ginsburg GS, West M, Harpole DH Jr, Nevins JR. A genomic strategy to refine prognosis in early-stage non-small-cell lung cancer. N Engl J Med. 2006 Aug 10;355(6):570-80. doi: 10.1056/NEJMoa060467. PMID 16899777 (Retraction: PMID 21366430 Potti A, Mukherjee S, Petersen R, Dressman HK, Bild A, Koontz J, Kratzke R, Watson MA, Kelley M, Ginsburg GS, West M, Harpole DH Jr, Nevins JR. N Engl J Med. 2011 Mar 24;364(12):1176)
- [Background] Potti A, Dressman HK, Bild A, Riedel RF, Chan G, Sayer R, Cragun J, Cottrill H, Kelley MJ, Petersen R, Harpole D, Marks J, Berchuck A, Ginsburg GS, Febbo P, Lancaster J, Nevins JR. Genomic signatures to guide the use of chemotherapeutics. Nat Med. 2006 Nov;12(11):1294-300. doi: 10.1038/nm1491. Epub 2006 Oct 22. PMID 17057710 (Retraction: PMID 21217686 Potti A, Dressman HK, Bild A, Riedel RF, Chan G, Sayer R, Cragun J, Cottrill H, Kelley MJ, Petersen R, Harpole D, Marks J, Berchuck A, Ginsburg GS, Febbo P, Lancaster J, Nevins JR. Nat Med. 2011 Jan;17(1):135)
- See also: Clinical Trials at Duke Cancer Institute — http://www.cancer.duke.edu/CTrials/index

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 31 patients were registered, but 7 patients were not assigned treatment due to genomic screening failure or study ineligibility. The remaining 24 patients were assigned to the vinorelbine and pemetrexed treatment arms.
Groups:
- Screen Failures: Patients who were registered and underwent protocol-based procedure (e.g. biopsy, genomic screening), but were not assigned to or administered genomics-directed, protocol-based therapy.
  Note that two patients who were assigned protocol-based treatment (1 in each arm) did not receive the treatment and were added to the 7 initially identified as screen failures within the summary of baseline characteristics and outcome measures.
Period: Overall Study
Arm/Group | Arm A-Vinorelbine | Arm B-Pemetrexed | Screen Failures
Started | 9 (Registered patients assigned to receive vinorelbine + cisplatin protocol therapy.) | 15 (Registered patients assigned to receive pemetrexed + cisplatin protocol therapy.) | 7 (Registered patients who were not assigned to receive protocol therapy.)
Assigned Treatment | 9 | 15 | 0
Completed | 8 (Patients who received vinorelbine + cisplatin protocol therapy.) | 14 (Patients who received pemetrexed + cisplatin protocol therapy.) | 0
Not Completed | 1 | 1 | 7
Not completed — Not Treated | 1 | 1 | 7

BASELINE CHARACTERISTICS:
Population: One patient in each of the vinorelbine and pemetrexed arms did not undergo protocol-based treatment, resulting in 22 total patients who were treated with either vinorelbine or pemetrexed. These two enrolled patients who were not administered treatment were added to the 7 original screen failures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A-Vinorelbine | Arm B-Pemetrexed | Screen Failures | Total
Number analyzed (Participants) | 8 | 14 | 9 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.13 (3.36) | 58.93 (9.14) | 61.44 (11.35) | 61.18 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 6 | 17
  Male | 5 | 6 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 8 | 14 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: 2-Year Progression-Free Survival Rate in Patients With Completely Resected Stage IB, II, or IIIA NSCLC
Description: Progression-free survival time was defined as the time from initiation of study treatment to the first date of disease progression or death as a result of any cause. Progression was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Time was censored at the date of the last follow-up visit for patients who were still alive and have not progressed. The two-year progression free survival rate is a percentage, representing the fraction of treated patients who, after two years, are disease free or alive.
Time Frame: 2 years
Population: Due to the irreproducible nature of the genomic signatures of chemotherapeutic sensitivity, analyses based on separate treatment groups were inappropriate. Therefore, all enrolled participants (initiated for treatment) from both treatment arms were analyzed together.
Measure: Number (95% Confidence Interval); unit: percentage of treated patients
Groups:
- Treatment: Treatment refers to patients treated in the combined vinorelbine and pemetrexed arms of the study. Due to the irreproducibility of the genomics-based prediction model for assigning patients into the original cisplatin treatment arms, patients from both arms were combined for primary outcome analysis.
Arm/Group | Treatment
Number analyzed (Participants) | 22
percentage of treated patients | 63.64 [40.29 to 79.88]

2. Secondary Outcome: Percentage of Patients With Completely Resected NSCLC Tumors That Can Be Analyzed and Used to Direct Adjuvant Chemotherapy
Description: The percentage of patients with completely resected NSCLC tumors who had successful genomic analysis and assigned to treatment among patients. All 31 patients enrolled in the study had completely resected tumors. These tumors included a mixture of squamous and non-squamous histologies as indicated the original protocol. However, an amendment dated January 25, 2010 limited eligibility to patients with non-squamous disease. Given that only 5 patients were accrued into the study after this amendment, results reported will consider all histologies.
Time Frame: 4 years
Measure: Number; unit: Percentage of participants
Groups:
- All Registered Patients: All registered/enrolled patients are included in this outcome, which was measured at the time of consent.
Arm/Group | All Registered Patients
Number analyzed (Participants) | 31
Percentage of participants | 77.4

3. Secondary Outcome: 2-Year Overall Survival in Patients Treated for NSCLC
Description: Overall survival time was defined as the time from initiation of study treatment to the date of death as a result of any cause. Time was censored at the date of the last follow-up visit for patients who were still alive. The two-year overall survival rate is a percentage, representing the fraction of treated patients who, after two years, are alive
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of treated patients
Groups:
- Treatment: Treatment refers to patients treated in the combined vinorelbine and pemetrexed arms of the study.
Arm/Group | Treatment
Number analyzed (Participants) | 22
percentage of treated patients | 81.81 [58.53 to 92.76]

4. Secondary Outcome: Patient Understanding and Perceptions of Participating in a Clinical Trial Evaluating Cancer Genomics for Adjuvant Treatment of Early Stage Lung Cancer
Description: Do to space limitations, see the Detailed Description in the study protocol for the wording of the questions used in the Patient Expectations Questionnaire.
Time Frame: Baseline
Population: Twenty-six questionnaires were returned. There was insufficient numbers to provide for substantive analysis.
Arm/Group | All Registered Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Compare Drug Sensitivity Patterns of Cisplatin and Pemetrexed in Both Treatment Arms
Description: Using genomics-based prediction models previously developed separately for cisplatin and pemetrexed, the probability that each patient was sensitive or would respond to treatment was computed. Quartiles describe the patterns of drug sensitivity probabilities. The 1st, 2nd, and 3rd quartiles are the sensitivity levels at which 25%, 50%, and 75% of patients have lower sensitivity. There is lack of integrity regarding the available data due to irreproducible genomic signatures. Therefore the results of this outcome are not presented.
Time Frame: 2 years
Population: There is lack of integrity regarding the available data due to irreproducible genomic signatures. Therefore the results of this outcome are not presented.
Arm/Group | Arm A-Vinorelbine | Arm B-Pemetrexed
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No adverse events were observed for patients considered screen failures.
Arm/Group | Arm A-Vinorelbine | Arm B-Pemetrexed
Serious Adverse Events (participants affected / at risk) | 4/8 | 2/14
Other Adverse Events (participants affected / at risk) | 8/8 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A-Vinorelbine (N=8) | Arm B-Pemetrexed (N=14)
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
General disorders and administration site conditions - Other, specify: Smell alteration (General disorders) | 1 | 0
Infections and infestations - Infection with Grade 3 or 4 neutrophils : Abdomen NOS (Infections and infestations) | 1 | 0
Infections and infestations - Infection with Grade 3 or 4 neutrophils: Blood (Infections and infestations) | 1 | 0
Infections and infestations - Infection with Grade 3 or 4 neutrophils: Lung (pneumonia) (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: Left interal carotid artery stenosis (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A-Vinorelbine (N=8) | Arm B-Pemetrexed (N=14)
Anemia (Blood and lymphatic system disorders) | 7 | 10
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specify: Tachycardia (Cardiac disorders) | 2 | 0
Ear and labyrinth disorders - Other, specify: vibrations and muffling (Ear and labyrinth disorders) | 0 | 2
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 9
Blurred vision (Eye disorders) | 1 | 3
Dry eye (Eye disorders) | 1 | 1
Eye disorders - Other, specify: Decreased visual acuity (Eye disorders) | 2 | 1
Watering eyes (Eye disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhea (Gastrointestinal disorders) | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorders - Other, specify: feeling of stomach fullness (Gastrointestinal disorders) | 1 | 2
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 6 | 11
Vomiting (Gastrointestinal disorders) | 1 | 5
Chills (General disorders) | 1 | 1
Edema face (General disorders) | 0 | 2
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 7 | 11
Fever (General disorders) | 1 | 1
General disorders and administration site conditions - Other, specify: Smell alteration (General disorders) | 0 | 1
Injection site reaction (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Immune system disorders - Other, specify: hives (Immune system disorders) | 0 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 1
Gum infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: infected cyst on neck (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Cholesterol high (Investigations) | 0 | 1
Creatinine increased (Investigations) | 4 | 3
Investigations - Other, specify: Decreased chloride (Investigations) | 6 | 4
Neutrophil count decreased (Investigations) | 6 | 9
Platelet count decreased (Investigations) | 2 | 2
Weight gain (Investigations) | 0 | 1
Weight loss (Investigations) | 3 | 2
White blood cell decreased (Investigations) | 5 | 5
Anorexia (Metabolism and nutrition disorders) | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatremia (Metabolism and nutrition disorders) | 6 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal and connective tissue disorder - Other, specify: Leg cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 6 | 5
Headache (Nervous system disorders) | 5 | 8
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: Left interal carotid artery stenosis (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 3
Urinary retention (Renal and urinary disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify: left base crackle/pleural rub (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3
Skin and subcutaneous tissue disorders - Other, specify: Chapped lips (Skin and subcutaneous tissue disorders) | 0 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No